CLINICAL TRIAL: NCT03885427
Title: Analgo-Sedative Effects Of Oral, Or Nebulized Ketamine In Pre-schoolers Undergoing Elective Surgery: A-Comparative Randomized Double Blind Study
Brief Title: Analgo-Sedative Effects Of Oral, Or Nebulized Ketamine In Pre-schoolers Undergoing Elective Surgery.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, Principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5296
Record Dates: First submitted 2019-03-14; First posted 2019-03-21 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Conscious Sedation; Postoperative Analgesia
Keywords: sedation; ketamine; analgesia; pre-schoolers
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: this will be a double blind study, and utilize a convenience sample of pre-schoolers. 31 children recruited in In oral ketamine arm, and 31 children in nebulized ketamine arm
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator will prepare the drug, and the out come assessor(the anesthesiologist not sharing in the study) will assess the primary, and secondary outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral ketamine (Experimental): evaluate sedative,and analgesic effects
  Interventions: Drug: Ketamine
- nebulized ketamine (Active Comparator): evaluate sedative, and analgesic effects
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — evaluate sedative, and analgesic effects of oral or nebulized ketamine
  Other Names: ketalar

SUMMARY:
the primary objective of this study is to investigate the sedative, and analgesic effects of oral, or nebulized ketamine as premedication drugs, and providing postoperative analgesia for the preschoolers and decrease their need for systemic analgesia.The secondary objective is to compare each sedation technique after oral, or nebulized ketamine for safety ,and procedural outcomes.

DETAILED DESCRIPTION:
Preoperative communication, premedication interventions, and being accompanied by parents are useful methods in decreasing preoperative separation anxiety , postoperative psychological trauma, and ensuring smooth induction for preschoolers undergoing elective surgery.

Procedural sedation, and analgesia was defined by O'Donnell as a drug induced state of decreasing awareness, pain, and memory that allowing patient continue his ,or her own protective reflexes, and moving purposefully( O' Donnell etal, 2003).

Ketamine is an anesthetic drug having sedative, and analgesic properties with different routes of administration in children (IV, intramuscular, subcutaneous, oral, rectal, sublingual, intranasal, and nebulized) .

Ketamine produces its analgesic properties in acut pain management from reversible antagonizing the N-methyl-D-aspartate (NMDA)receptors , reducing levels of many proinflammatory mediators in the acute phase, and acting on other non-NMDA pathways that playing important roles in pain, and mood regulation, like its effect on µ-opioid receptors, nicotinic, muscarinic cholinergic, ɣ-aminobutyric acid receptors, activation of high -affinity D2 dopamine receptors, and L-type voltage-gated calcium channels.

The oral route is the most popular than other routes ,as it's safe, efficient, acceptable, and familiar for pediatric patients..

Oral ketamine often requires higher, and frequent doses as it's bioavailability is lower (17-24%) compared to IV (100%),Intramuscular (93%), sublingual/transbuccal(30%), intranasal(25-50%),and inhaler (70%) due to extensive first pass metabolism in liver, and intestine.

Ketamine inhalation is safe, rapid absorption, and affordable route of administration.

ELIGIBILITY:
Inclusion Criteria:

* Parents acceptance.
* Age (3-6) years old.
* American Society of Anesthesiologist physical status (ASA) I / II
* Elective surgery of approximately half to one hour duration under general anesthesia.
* Child With Body Mass Index (BMI) (15-18kg/m²)

Exclusion Criteria:

* Parents refusal.
* Altered mental status, and epilepsy.
* History of allergy to ketamine.
* Recent respiratory tract infection.
* Sever dysfunction of the central nervous system.
* Increased intracranial pressure, and increased intra-ocular pressure.
* Cardiac dysrhythmia ,and/or congenital heart disease.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
evaluate sedative effects of oral, or nebulized ketamine in preschoolers undergoing elective surgery | 30 minutes.
  • To assess onset time of sedation by sedation scale (SS-5) score.
  The sedation scale:
  1. Rarely awake, needs shaking, or shouting to wake up.
  2. Asleep, eyes closed, wake up when called softly,or lightly touched.
  3. Sleepy, but eyes open spontaneously.
  4. Awake.
  5. Agitated.
compare each sedation technique for the time of separation state. | at 30 minutes after drug intake
  The separation state will be assessed and designated as satisfactory separation if the Emotional State Scale (ESS-4) score will be no more than two points.
  The Emotional State Scale (ESS-4):
  1. Calm.
  2. Apprehensive, not smiling, tentative behavior, withdrawn.
  3. Crying.
  4. Thrashing, crying with movements of the arms, and legs, resisting.
compare the sedation technique for successful venous cannulation. | at time of attempted cannulation, regardless of whether the vein is actually cannulated on the first attempt.
  Successful venous cannulation is defined as an Emotional State Scale (ESS-4≤ 2).
  The Emotional State Scale (ESS-4):
  1. Calm.
  2. Apprehensive, not smiling, tentative behavior, withdrawn.
  3. Crying.
  4. Thrashing, crying with movements of the arms, and legs, resisting.

SECONDARY OUTCOMES:
to compare the intensity of pain postoperative. | immediately after recovery, and every half hour for four hours postoperative
  the intensity of pain will be assessed using modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS).
  Score 1 2 3 Cry No cry Crying, moaning Scream Facial Smiling Composed Grimace Verbal Positive None, or other complaints Pain complaint Torso Neutral Shifting, tense, upright Restrained Leg Neutral kicks, squirm, drawn up Restrained Touch No touching Reach, touch, grab Restrained CHEOPS pain score=SUM(0)(points for all 6 parameters). Interpretation : minimum score:6, maximum score:18.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University Hospitsals, Zagazig, Egypt